CLINICAL TRIAL: NCT00134095
Title: Phase II Clinical Study of Preoperative S-1/CPT-11 Combination Chemotherapy in Patients With Locally Advanced Gastric Cancer
Brief Title: S-1 and Irinotecan in Treating Patients Who Are Undergoing Surgery for Locally Advanced Stomach Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fukushima Medical University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000439474; FMUH-UHA-GC04-02
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2010-01

CONDITIONS: Gastric Cancer
Keywords: adenocarcinoma of the stomach; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: tegafur-gimeracil-oteracil potassium
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as S-1 and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy before surgery may shrink the tumor so that it can be completely removed.

PURPOSE: This phase II trial is studying how well giving S-1 together with irinotecan works in treating patients who are undergoing surgery for locally advanced stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of neoadjuvant S-1 and irinotecan in patients with locally advanced gastric cancer.

Secondary

* Determine the histological response in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine postoperative morbidity in patients treated with this regimen.
* Determine the rate of potentially curative surgery in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral S-1 on days 1-21 and irinotecan IV over 90 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo gastrectomy with lymphadenectomy. After surgery, patients resume treatment with S-1 alone as before for 1 year.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric adenocarcinoma

  * Locally advanced disease

    * Clinical stage T3-4, N0-3, M0 (according to the Japanese gastric cancer classification)
* Planning to undergo curative surgery after neoadjuvant chemotherapy

PATIENT CHARACTERISTICS:

Age

* 20 to 75

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC 4,000-12,000/mm^3
* Granulocyte count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* AST and ALT ≤ 100 U/L
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 50 mL/min

Pulmonary

* PaO_2 > 60 mm Hg on room air

Other

* Able to swallow oral medication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for gastric cancer

Chemotherapy

* No prior chemotherapy for gastric cancer

Endocrine therapy

* No prior endocrine therapy for gastric cancer

Radiotherapy

* No prior radiotherapy for gastric cancer

Surgery

* No prior surgery for gastric cancer

Other

* No other prior therapy for gastric cancer

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Tumor shrinkage
Historical tumor shrinkage
Overall survival
Progression-free survival
Median survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Mitsukazu Gotoh, MD, Study Chair — Fukushima Medical University Hospital
Locations (7):
- Japan (7):
  - Yamamoto Kumiai General Hospital, Noshiro, Akita
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Asahikawa Kosei General Hospital, Asahikawa, Hokkaido
  - Kobe City General Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tsuruoka Municipal Shonai Hospital, Tsuruoka, Yamagata
  - Yamagata Prefectural Central Hospital, Yamagata, Yamagata